CLINICAL TRIAL: NCT00876200
Title: The Efficacy of Minoxidil in Children With Williams-Beuren Syndrome: a Randomized Clinical Trial.
Brief Title: Efficacy of Minoxidil in Children With Williams-Beuren Syndrome
Acronym: Williams
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006.437/30
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2016-01

CONDITIONS: Williams Beuren Syndrome
Keywords: Williams Beuren syndrome; Cardiovascular abnormalities; Cardiovascular structure
MeSH Terms: conditions — Williams Syndrome; Cardiovascular Abnormalities | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minoxidil (Experimental): Normotension: 0.2mg/kg/day for children under 12 and 5mg/day for children aged 12 or more.
  Hypertension: 0.2mg/kg/day, increasing up to a maximal dosage of 1 mg/kg) for children under 12. 5mg/day, increasing as needed of 0.1 mg/kg/day (up to a maximal dosage of 40 mg/day) for children aged 12 or more.
  Interventions: Drug: Minoxidil
- Placebo (Placebo Comparator): Placebo = lactose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minoxidil — Normotension: 0.2mg/kg/day for children under 12 and 5mg/day for children aged 12 or more.
  Hypertension: 0.2mg/kg/day, increasing up to a maximal dosage of 1 mg/kg) for children under 12. 5mg/day, increasing as needed of 0.1 mg/kg/day (up to a maximal dosage of 40 mg/day) for children aged 12 or more.
  Arms: Minoxidil
Drug: Placebo — Normotension: 0.2mg/kg/day for children under 12 and 5mg/day for children aged 12 or more.
  Hypertension: 0.2mg/kg/day, increasing up to a maximal dosage of 1 mg/kg) for children under 12. 5mg/day, increasing as needed of 0.1 mg/kg/day (up to a maximal dosage of 40 mg/day) for children aged 12 or more.
  Arms: Placebo

SUMMARY:
The Williams-Beuren syndrome (WBS) is a sporadic congenital disorder characterized by a multisystem developmental impairment. This syndrome is caused by a microdeletion in chromosome 7q11.23 that encompasses loss of the elastin locus.

Elastin, which is part of the extracellular matrix, controls proliferation of vascular smooth muscle cells (VSMCs) and stabilizes arterial structure. Loss of elastin gene in WBS patients has been claimed to provide a biological basis for the abnormal elastic fibre properties leading to cardiovascular abnormalities like supravalvular aortic stenosis (SVAS), hypertension, arteriosclerosis and stenosis in more than 50% of WBS children.

These cardiovascular pathologies result in important consequences and neither curative nor preventive medicinal treatments exist at this time. Surgery is needed in more than half cases, while it is often leading to complications.

Minoxidil is a well-known antihypertensive drug used in adults and children. Furthermore, according to animal studies, minoxidil seems to increase arterial elastin content by decreasing elastase activity in these tissues. Other data demonstrate that minoxidil specifically stimulate elastin synthesis.

Working Hypothesis:If insufficient elastin synthesis leads to vascular complications and arterial hypertension in children with WBS, restoration of sufficient quantity of elastin should then result in prevention or inhibition of vascular malformations and improvement in arterial tension. Therefore, as a pharmacological agent capable to stimulate elastin expression, minoxidil might be a useful drug for the treatment of abnormal elastin metabolism in WBS children.

Objective:To evaluate the efficacy of minoxidil on cardiovascular structure in children with Williams Beuren syndrome.

Methodology: randomized controlled trial on two parallel group (23 patients in each arm) Main criterion:variation of carotid Intima-media thickness (IMT) before and after 12 months of treatment with Minoxidil versus placebo Secondary intermediate criteria of the vascular properties are arterial stiffness, cardiac and renal stenosis, arterial tension.

Total study duration:30 months including a 12 month-recruitment period

ELIGIBILITY:
Inclusion Criteria:

* proven diagnosis of Williams Beuren syndrome (genetic test)
* normotension or hypertension, treated or not
* male or female,
* 6< age <18,
* negative pregnancy test for childbearing potential female
* effective birth control for sexually active female
* signed consent form collected from parents or legal guardian

Exclusion Criteria:

* pulmonary hypertension secondary to mitral stenosis
* myocardial infarction within 1 month prior randomization
* known allergies to minoxidil or any of the components of Lonoten.
* asthma
* renal failure (creatinine clearance <40ml/min)
* no affiliation to a national health insurance program (social security)
* intolerance to lactose
* current vasodilator anti hypertensive treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2009-03; Primary Completion 2015-02 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Behrouz KASSAI, MD, Principal Investigator — Hospices Civils de Lyon
Locations (18):
- France (18):
  - Service de Cardiologie Pédiatrique, CHU Angers, Angers
  - Service de Cardiologie, Hôpital Saint-André, CHU Bordeaux, Bordeaux
  - Service de Néphrologie Pédiatrique, Hôpital Pellegrin, CHU Bordeaux, Bordeaux
  - Service de Génétique Médicale, Hôpital Pellegrin, CHU Bordeaux, Bordeaux
  - Département de Pédiatrie, Hôpital Femme Mère Enfant, Bron
  - Service de Cardiologie Pédiatrique, Hôpital Cardiovasculaire L. Pradel, Bron
  - Service Cardiologie, CHU St Jacques, Clermont-Ferrand
  - Département de Pédiatrie- Service de Cardiologie, CHU Grenoble, Grenoble
  - Service de Néphrologie Pédiatrique, CHRU de Lille, Lille
  - Service des Maladies Cardiovasculaires Infantiles et Congénitales, CHRU Lille, Lille
  - Service de Cardiologie Infantile, CHU Nancy, Nancy
  - Service de Cardiologie Pédiatrique, Hôpital Necker Enfants Malades, Paris
  - Service de Physiologie, Explorations Fonctionnelles, Hôpital Robert Debré, Paris
  - Unité de Pharmacologie Clinique, Hôpital Robert Debré, Paris
  - Service de Pathologie Cardiaque Congénitale du Fœtus, de l'Enfant et de l'Adulte, Hôpital Haut Lévêque, CHU de Bordeaux, Pessac
  - Service de Génétique Médicale, CHU La Milétrie, Poitiers
  - Service de Cardiologie - Hôpital des Enfants, Toulouse
  - Service de Néphrologie Pédiatrique - Hôpital des Enfants, CHU Toulouse, Toulouse

REFERENCES:
- [Result] Kassai B, Bouye P, Gilbert-Dussardier B, Godart F, Thambo JB, Rossi M, Cochat P, Chirossel P, Luong S, Serusclat A, Canterino I, Mercier C, Rabilloud M, Pivot C, Pirot F, Ginhoux T, Coopman S, Grenet G, Gueyffier F, Di-Fillippo S, Bertholet-Thomas A. Minoxidil versus placebo in the treatment of arterial wall hypertrophy in children with Williams Beuren Syndrome: a randomized controlled trial. BMC Pediatr. 2019 May 28;19(1):170. doi: 10.1186/s12887-019-1544-1. PMID 31138170
- See also: Related Info — http://www.autourdeswilliams.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Minoxidil: Normotension: 0.2mg/kg/day for children under 12 and 5mg/day for children aged 12 or more.
  Hypertension: 0.2mg/kg/day, increasing up to a maximal dosage of 1 mg/kg) for children under 12. 5mg/day, increasing as needed of 0.1 mg/kg/day (up to a maximal dosage of 40 mg/day) for children aged 12 or more.
  Minoxidil: Normotension: 0.2mg/kg/day for children under 12 and 5mg/day for children aged 12 or more.
  Hypertension: 0.2mg/kg/day, increasing up to a maximal dosage of 1 mg/kg) for children under 12. 5mg/day, increasing as needed of 0.1 mg/kg/day (up to a maximal dosage of 40 mg/day) for children aged 12 or more.
- Placebo: Placebo = lactose
  Placebo: Normotension: 0.2mg/kg/day for children under 12 and 5mg/day for children aged 12 or more.
  Hypertension: 0.2mg/kg/day, increasing up to a maximal dosage of 1 mg/kg) for children under 12. 5mg/day, increasing as needed of 0.1 mg/kg/day (up to a maximal dosage of 40 mg/day) for children aged 12 or more.
Period: Overall Study
Arm/Group | Minoxidil | Placebo
Started | 9 | 12
Completed | 8 | 9
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minoxidil | Placebo | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.33 (4.42) | 10.75 (3.77) | 11.43 (4.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 4 | 8 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History of hypertension [Count of Participants; unit: Participants] | 2 | 2 | 4
History of cardiovascular disease [Count of Participants; unit: Participants] | 4 | 6 | 10
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 128.11 (16.78) | 120.83 (12.68) | 123.95 (14.65)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.22 (15.58) | 73.17 (8.97) | 75.33 (12.16)
BMI [Mean (Standard Deviation); unit: Kg/cm2] | 17.93 (3.88) | 17.54 (3.30) | 17.71 (3.47)

OUTCOME MEASURES:

1. Primary Outcome: Variation of Carotid Intima-media Thickness (IMT) Assessed by Vascular Echography
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Minoxidil | Placebo
Number analyzed (Participants) | 9 | 9
mm | 0.028 [0.002 to 0.058] | 0.012 [0.0017 to 0.040]

2. Secondary Outcome: Efficacy of Minoxidil on Humeral IMT Assessed by Vascular Echography
Time Frame: 18 months
Reporting Status: Not Posted

3. Secondary Outcome: Efficacy of Minoxidil on Arterial Stiffness (Pulse Wave Velocity and Vascular Compliance at J0, M12 and M18)
Time Frame: 18 months
Reporting Status: Not Posted

4. Secondary Outcome: Efficacy of Minoxidil on Supravalvular Stenosis, Pulmonary Stenosis, Aortic Stenosis and Renal Stenosis (Cardiac and Renal Echodoppler at J0, and M12)
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Efficacy of Minoxidil on Arterial Tension (24H-Holter at J0 and M12)
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Effect of Minoxidil on Neurohumoral Mechanisms of Cardiovascular Regulation and on Plasmatic Markers of the Extracellular Matrix.
Time Frame: 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Genetic Study: Characterization of Deletions Responsible for WBS (Size Deletion, DNA Sample at Inclusion).
Time Frame: Day 0
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Minoxidil | Placebo
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/12
Other Adverse Events (participants affected / at risk) | 5/9 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minoxidil (N=9) | Placebo (N=12)
Flat foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Strabismus correction (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minoxidil (N=9) | Placebo (N=12)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes